CLINICAL TRIAL: NCT06413290
Title: Doppler Evaluation of Ultrasound-guided Pectointercostal Fascial Plane Block in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18/12
Record Dates: First submitted 2024-04-24; First posted 2024-05-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Surgery
Keywords: regional anesthesia; postoperative pain; doppler ultrasound; cardiovascular surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PIFP block group: Before the anesthesia induction, PIFP block will be performed
  Interventions: Other: PIFP block group
- Control group: No intervention
  Interventions: Other: Control group

INTERVENTIONS:
Other: PIFP block group — Ultrasound-guided PIFP block will be performed approximately 30 minutes before surgery in patients undergoing cardiac surgery
  Groups: PIFP block group
Other: Control group — No intervention
  Groups: Control group

SUMMARY:
The aim of this study was to evaluate the effect of pectointercostal fascial plane block on regional haemodynamic parameters in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Perioperative pain management has become an important component of Enhanced Recovery After Surgery (ERAS) protocols in patients undergoing cardiac surgery. Pain is most intense in the first two days after cardiac surgery. Inadequate pain control has been shown to cause an increase in pulmonary complications due to inadequate mobility and coughing, an increase in sympathetic activation, an increase in myocardial infarction and thromboembolic events, delayed wound healing, and prolonged hospital and intensive care unit stay. Non-steroidal anti-inflammatory drugs (NSAIDs), paracetamol, opioids, epidural anesthesia and ultrasound-guided fascial plane blocks are widely used for pain management after cardiac surgery. The pectointercostal fascial plane (PIFP) block is an ultrasound-guided, superficial fascial plane block that can be applied as part of multimodal postoperative analgesia, especially after cardiac surgery. PIFB block has been shown to reduce postoperative analgesic consumption and improve pain scores not only in patients undergoing cardiac surgery but also in non-cardiac surgeries and thoracic procedures. The aim of this study was to evaluate the effect of PIFP block on regional haemodynamic parameters in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery
* over 18 years, adult
* American Society of Anaesthesiology (ASA) I-III

Exclusion Criteria:

* history of cerebrovascular disease
* history of Alzheimer's disease
* mental disorder
* emergency surgery
* re-operated due to surgery-related complications
* allergy to local anaesthetics
* declining to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include ASA I-III adult patients who are planned to undergo elective cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
blood volume | 1 hour
  The regional haemodynamic impact of PIDB block will be evaluated by Doppler ultrasound

SECONDARY OUTCOMES:
postoperative opioid consumption | 24 hours
  The amount of postoperative opioid consumption will be recorded
postoperative Numerical Rating Scale (NRS) pain scores | 24 hours
  The postoperative pain intensity will be assessed with NRS pain scores (0=no pain, 10=worst possible pain)
length of hospital stay | 5 days
  The interval from the end of the surgery until the patient's discharge will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu O Karaveli, M.D., Study Director — University of Health Sciences, Antalya Training and Researh Hospital
Locations (1):
- University of Health Sciences, Antalya Training and Research Hospital, Antalya, Muratpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khera T, Murugappan KR, Leibowitz A, Bareli N, Shankar P, Gilleland S, Wilson K, Oren-Grinberg A, Novack V, Venkatachalam S, Rangasamy V, Subramaniam B. Ultrasound-Guided Pecto-Intercostal Fascial Block for Postoperative Pain Management in Cardiac Surgery: A Prospective, Randomized, Placebo-Controlled Trial. J Cardiothorac Vasc Anesth. 2021 Mar;35(3):896-903. doi: 10.1053/j.jvca.2020.07.058. Epub 2020 Jul 24. PMID 32798172
- [Background] Ata F, Yilmaz C. Retrospective Evaluation of Fascial Plane Blocks in Cardiac Surgery With Median Sternotomy in a Tertiary Hospital. Cureus. 2023 Mar 3;15(3):e35718. doi: 10.7759/cureus.35718. eCollection 2023 Mar. PMID 37016643